CLINICAL TRIAL: NCT07376239
Title: Quality of Life, Depression and Sexual Function in Men Living With HIV Under Effective Antiretroviral Therapy Compared With Healthy Controls
Brief Title: Quality of Life, Depression and Sexual Function in Men Living With HIV
Status: Enrolling by invitation | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Özlem Güler, Assistant Professor M.D., Kocaeli University
Other Study IDs: GOKAEK-2025/19/06 2025/450
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: HIV Infections
Keywords: HAART; Sustained virologic response; Health surveys; Psychological wellbeing; Sexual health
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men living with HIV: Heterosexual adult men with HIV receiving combination antiretroviral therapy and with confirmed virologic suppression who complete quality-of-life, depression, and sexual-function questionnaires.
- Healthy controls: HIV-negative adult men without major medical conditions who complete the same quality-of-life, depression, and sexual-function questionnaires for comparison.

SUMMARY:
This observational case-control study evaluates quality of life, depressive symptoms, and sexual function in heterosexual men living with HIV who are receiving effective combination antiretroviral therapy and have achieved virologic suppression, compared with healthy male controls. Participants complete validated questionnaires assessing quality of life (EUROHIS-QOL-8), depression (Beck Depression Inventory), and sexual function (Arizona Sexual Experience Scale). The study aims to identify psychosocial and sexual health challenges that may persist despite effective HIV treatment.

DETAILED DESCRIPTION:
Combination antiretroviral therapy (cART) has markedly improved survival and virologic outcomes in people living with HIV; however, impairments in quality of life, mental health, and sexual function may persist even under long-term effective treatment. These outcomes are clinically important because they influence treatment adherence, overall wellbeing, and long-term health.

This is a comparative, observational, case-control study conducted at the outpatient clinic of the Department of Infectious Diseases and Clinical Microbiology at Kocaeli University Hospital. The study includes heterosexual men living with HIV who are receiving regular cART and have achieved virologic suppression confirmed at two consecutive visits. A control group of healthy male volunteers matched for age and key sociodemographic characteristics is recruited from companions of patients attending the same clinic.

During a three-week recruitment period, all eligible participants are invited to complete a set of validated self-report questionnaires in a quiet environment without researcher interference. Sociodemographic data are collected, including age, educational status, marital status, physical activity, living conditions, smoking, and alcohol use.

Quality of life is assessed using the EUROHIS-QOL-8 (WHOQOL-8), depressive symptoms are measured using the Beck Depression Inventory (BDI), and sexual function is evaluated using the Arizona Sexual Experience Scale (ASEX), all of which have validated Turkish versions. These instruments provide continuous measures of wellbeing, depression severity, and sexual dysfunction.

The primary objective is to compare quality of life, depression, and sexual function between men living with HIV and healthy controls. Secondary objectives include evaluating correlations between depression, sexual function, quality of life, and age within each group. The results are intended to clarify the psychosocial and sexual health burden among virologically suppressed men living with HIV and to inform routine screening and supportive care strategies in HIV clinics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Male sex
* Heterosexual orientation
* Confirmed diagnosis of HIV infection
* Receiving combination antiretroviral therapy (cART)
* Virologic suppression confirmed at two consecutive visits
* Ability to understand and complete the questionnaires

Exclusion Criteria:

* Female sex
* Age < 18 years
* Advanced HIV disease
* Presence of significant comorbid medical conditions
* Cognitive impairment or communication difficulties that could interfere with completion of the survey

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group consisted of heterosexual men living with HIV (MLWH) who were receiving cART and had achieved virological suppression, confirmed at least at two separate visits. The control group comprised volunteers among the companions of patients attending the same clinic for other medical reasons, who were matched for age and basic demographic characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life score (EUROHIS-QOL-8) | Baseline (at study enrollment; single assessment)
  Quality of life measured using the EUROHIS-QOL-8 questionnaire. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Depression severity (Beck Depression Inventory) | Baseline (at study enrollment; single assessment)
  Depressive symptoms measured using the Beck Depression Inventory (BDI). Higher scores indicate more severe depression.
Sexual function (Arizona Sexual Experience Scale) | Baseline (at study enrollment; single assessment)
  Sexual function measured using the Arizona Sexual Experience Scale (ASEX). Higher scores indicate greater sexual dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Güler, MD, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided